CLINICAL TRIAL: NCT03148093
Title: The CHOICE Registry: A Research Initiative Examining Clinical, Economic, and Humanistic Outcomes in the Management of Metastatic Colorectal Cancer
Brief Title: The CHOICE Registry
Status: Terminated | Type: Observational
Why Stopped: Competing clinical trials and slower than expected patient enrollment
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-102-01
Record Dates: First submitted 2017-04-04; First posted 2017-05-10 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Registry; Patient Reported Outcomes; Treatment Patterns; Prescription Use
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CHOICE Registry will describe real-world treatment patterns and physician and patient (and caregiver)-reported outcomes associated with patients who have progressed beyond 2nd line metastatic colorectal cancer.

DETAILED DESCRIPTION:
A prospective, non-interventional, observational, approach will be employed. All patient follow-up visits and other interactions will be established by the physician investigator: the CHOICE Registry will not impose a fixed schedule of follow-up visits. Data will be obtained in conjunction with actual follow-up visits to support treatment and various assessments of disease progression, patient quality of life and caregiver burden, and resource utilization. Patients will be followed for minimum of 15 months. All prescribed and administered medications, treatment adjustments and duration will be documented by the physician investigator treating the patient as per standard of care. The CHOICE Registry will not impose any change to the treatment regimen prescribed by physicians participating in the Registry. Adult males and females with metastatic colorectal cancer (having received first and second line treatment, and upon initiation of third line or later treatment) will be eligible to participate. Approximately 1000 patients will be enrolled by approximately 30 to 40 physician investigators representing both community and academic medical centers in the United States. Descriptive statistics will be employed to address the key research objectives of the CHOICE Registry, such as a description of patients receiving various second (and/or subsequent) lines of treatment in the management of metastatic colorectal cancer in real world clinical settings, and the associated clinical, economic, and humanistic (patient-reported) outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Diagnosis of metastatic CRC
3. Having completed first and second lines of treatment for metastatic CRC
4. Intending (at time of enrollment) to initiate a third (or subsequent) line of treatment
5. Ability to understand and read English or Spanish
6. Willing and able to sign an Informed Consent Form (ICF), or have a Legally Authorized Representative willing and able to consent on the patient's behalf

Exclusion Criteria:

1. Patient is unwilling or unable to participate in the Registry at the time of enrollment
2. The patient is currently participating in an investigational clinical trial
3. Patients not having mental capacity and or ability to participate in the Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from community and academic medical centers in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Real-world treatment patterns as assessed by FACT/NCCN-Colorectal Symptom Index-19 (FCSI-19) | Approximately 15 months
Real-world treatment patterns as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Approximately 15 months
Real-world treatment patterns as assessed by EuroQoL EQ-5D-5L | Approximately 15 months
Real-world treatment patterns as assessed by Medication Satisfaction Questionnaire (MSQ) | Approximately 15 months
Real-world treatment patterns as assessed by Modified Caregiver Strain Index (MCSI) | Approximately 15 months
Real-world treatment patterns as assessed by Work Productivity and Activity Impairment - Caregiver (WPAI) | Approximately 15 months
Real-world treatment patterns as assessed by Healthcare resource utilization (physician visits, pharmacotherapy, hospitalizations, etc.) | Approximately 15 months
Duration of therapy | Approximately 15 months
Reasons for dose adjustments and/or discontinuation of treatments | Approximately 15 months

SECONDARY OUTCOMES:
Healthcare Resource Utilization | Approximately 15 months
  To characterize (physician visits, pharmacotherapy, hospitalizations, etc.) in patients receiving various treatment regimens
Quality-of-life of patients receiving specific treatment regimens for mCRC per FACT/NCCN-Colorectal Symptom Index-19 (FCSI-19) | Approximately 15 months
Quality-of-life of patients receiving specific treatment regimens for mCRC per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Approximately 15 months
Utility of patients receiving specific treatment regimens for mCRC per EuroQoL EQ-5D-5L | Approximately 15 months
Treatment satisfaction in patients receiving various treatment regimens for mCRC per Medication Satisfaction Questionnaire (MSQ) | Approximately 15 months
Burden for caregivers providing support to patients enrolled in the registry per Modified Caregiver Strain Index (MCSI) | Approximately 15 months

OTHER OUTCOMES:
Overall Survival | Approximately 15 months
  Overall survival is defined as the time from the date of randomization to the date of death
Progression free survival | Approximately 15 months
  Progression free survival is defined as the time from the date of randomization until radiological disease

CONTACTS AND LOCATIONS:
Locations (1):
- Ingalls Memorial Hospital, Harvey, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided